CLINICAL TRIAL: NCT04734951
Title: Effect of a Power/Resistance Exercise Program and Oral Supplementation With Beta-hydroxy-beta-methyl Butyrate (HMB) on the Muscle Quality Index in Older Adults. A Randomized Controlled Trial
Brief Title: Muscle Quality Index Improvement by Exercise and HMB Oral Supplementation in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Responsible Party: Principal Investigator, Ariadna del Villar Morales, Medical Specialist in Physical Activity and Sports Medicine, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 34/20
Record Dates: First submitted 2020-12-14; First posted 2021-02-02 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Aging Well
Keywords: Older Adults; Muscle quality index; Exercise training; HMB

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power/resistance exercise (Active Comparator): Participants on a power/resistance exercise program
  Interventions: Other: Power/resistance exercise program
- Power/resistance exercise + HMB (Experimental): Participants on combined power/resistance exercise program + HMB oral supplementation
  Interventions: Other: Power/resistance exercise program; Dietary Supplement: HMB supplementation

INTERVENTIONS:
Other: Power/resistance exercise program — participants will complete a power/resistance program during 14 weeks. The exercise program will consist of training to improve muscle strength, neuromotor skills, flexibility, endurance, and a greater emphasis on maximum strength and power. The intensity will be set according the estimated repetition to failure.
Dietary Supplement: HMB supplementation — Daily oral supplementation with 237 ml of a polymeric nutritional formula added with 1.5 g of HMB (Ensure Advance®)
  Arms: Power/resistance exercise + HMB

SUMMARY:
The aging process is accompanied by a decrease in several biological and physical functions, which have an impact on the perception of well-being and quality of life. Among these, the decrease in muscle mass, strength and power are of particular importance as they are associated with poor cardiorespiratory function, functional limitations and mortality. The muscle quality index (MQI) is considered a key determinant of muscle function in adulthood. The main treatment to preserve muscle mass has been strength exercise and in some cases the use of aids that influence protein metabolism such as beta-hydroxy-beta-methyl butyrate (HMB), but the evidence on this topic is not consistent and is inconclusive. Therefore, the main purpose of this study is to investigate if the combination of a power/resistance exercise program and oral supplementation with HMB can improve the quality mass index in adults aged compared with those received a single exercise program after 14 weeks of intervention.

DETAILED DESCRIPTION:
Study design: this is a 14-week, randomized controlled trial. 76 participants will be recruited from the medical services of the National Institute of Rehabilitation (NIR).

Participants: Adults between 65-75 years old, with a body mass index between 25-30 kg/m^2, sedentaries, non-smokers, with compensated comorbidities, and who do not consume nutritional supplements will be recruited. Participants with uncompensated metabolic diseases, with high risk of falls (evaluated with Tinetti scale), frailty syndrome, and b2-adrenergic agonists, glucocorticoids, diuretics or peripheral vasodilators users will not be recruited.

Intervention: Participants will be randomized to 1) power/resistance exercise program (GEx), 2) power/resistance exercise program + HMB group (GExHMB) with computer-generated random numbers. The exercise program will consist of training to improve muscular strength, neuromotor skills, flexibility, endurance, and a greater emphasis on maximum strength and power. Every training session will consist of 15 minutes of warm-up, 40 to 60 minutes of power/resistance training, neuromuscular and aerobic exercises, and 15 minutes of cool-down. The power/resistance and neuromuscular training will be performed 3 days/week, 2-5 sets, 5-15 repetitions for each exercise according to the recommendation of the American College of Sports Medicine training progression models; the aerobic exercise will be performed 2 days/week. All exercises will be performed at moderate intensity and will take place in the NIR Sports Medicine therapeutic gym.

Oral supplementation with HMB will be from a commercial polymeric formula in liquid form (Ensure Advanced®, 230 ml); the supplement intake will be 1 bottle/day. All patients, regardless of the intervention, will be monitored by sports medicine physicians and nutritionists in order to promote adherence to treatment.

The muscle quality index (MQI) will be obtained from the determination of muscular strength by isokinetic dynamometry (at 60°/s) for the lower extremities and by hand dynamometry for the upper extremities; the lean segmental mass in the upper and lower extremities will be determined by 3-frequency electronic bioimpedance analysis. The MQI will be calculated from the muscular strength divided by the muscular mass.

Lower extremities muscular power will be determined by isokinetic dynamometry at 180°/s, physical performance will be assessed by the Short Physical Performance battery (SPPB) and quality of life perception will be evaluated by the EuroQoL-5D questionnaire. As part of the safety measures for the participants, liver function will be monitored by laboratory tests (liver enzyme profile and general urine test) which will be performed at the NIR laboratory.

For each participant the study length will be 14 weeks with 61 exercise sessions for the GEx and GExHMB groups and 98 days of oral supplementation for the GExHMB group. The beginning of the study corresponds to session 1 of exercise and day 1 of supplementation intake. Initial evaluations will be performed 5 days prior to the start of the intervention, while final evaluations will be conducted at the end of 14 weeks of follow-up (2 days after the last day of the intervention). Data will be recorded by study investigators blinded to participant assignment.

Comparison: Comparison group will receive the unique intervention of a strength/resistance exercise program.

Outcomes: The primary outcome is the upper and lower extremities MQI mean change. The secondary outcomes are mean changes in muscular power, physical performance, and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 25-30 km/m^2
* Appendicular skeletal muscle mass index in women ≥ 5.0 kg/m^2 and men ≥ 6.0 kg/m^2
* No regular exercise
* Non-smokers
* Compensated comorbidities
* Without consumption of nutritional supplements

Exclusion Criteria:

* Osteoporosis
* Cardiovascular diseases (recent heart attack, unstable angina, heart failure, complete atrioventricular block)
* Musculoskeletal injuries
* Severe cognitive impairment
* Major depressive disorder
* Thyroid diseases
* Anemia with no response to previous treatment in the last 3 months
* b2-adrenergic agonists, glucocorticoids, diuretics or peripheral vasodilators users
* With amino acid and vitamin D supplementation or suspended with less than 3 months
* Data of renal insufficiency
* Chronic obstructive pulmonary disease
* Malabsorption syndrome associated with malnutrition
* High risk of falls evaluated with the Tinetti scale (score ≤19)
* Frailty syndrome

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline arm Muscle Quality Index (MQIarm) | Baseline and 14 weeks
  The muscle quality index from dominant arm will be calculated with data obtained from hand grip strength, and lean mass obtained by bioimpedance analysis according with the formula:
  MQIarm = hand grip strength (kg) / arm lean mass (kg)
Mean change from baseline leg Muscle Quality Index (MQIleg) | Baseline and 14 weeks
  The muscle quality index from dominant leg will be calculated with data obtained by isokinetic, and lean mass obtained by bioimpedance analysis according with the formula:
  MQIleg = peak torque (Nm) / leg lean mass (kg)

SECONDARY OUTCOMES:
Mean change from baseline muscular power | Baseline and 14 weeks
  The muscular power will be determined by isokinetic dynamometry at 180°/s
Short Physical Performance Battery (SPPB) | Baseline and 14 weeks
  Short Physical Performance Battery scale, range 0-12. The higher the score, the better the physical performance
Health-related quality of life | Baseline and 14 weeks
  EuroQol-5D (5 dimension) scale; the lower the level (1-3), the better the health state

CONTACTS AND LOCATIONS:
Overall Officials: Ariadna d Morales, MD, Principal Investigator — National Institute of Rehabilitation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fragala MS, Kenny AM, Kuchel GA. Muscle quality in aging: a multi-dimensional approach to muscle functioning with applications for treatment. Sports Med. 2015 May;45(5):641-58. doi: 10.1007/s40279-015-0305-z. PMID 25655372
- [Background] Barbieri E, Agostini D, Polidori E, Potenza L, Guescini M, Lucertini F, Annibalini G, Stocchi L, De Santi M, Stocchi V. The pleiotropic effect of physical exercise on mitochondrial dynamics in aging skeletal muscle. Oxid Med Cell Longev. 2015;2015:917085. doi: 10.1155/2015/917085. Epub 2015 Apr 5. PMID 25945152
- [Background] Barbat-Artigas S, Rolland Y, Zamboni M, Aubertin-Leheudre M. How to assess functional status: a new muscle quality index. J Nutr Health Aging. 2012 Jan;16(1):67-77. doi: 10.1007/s12603-012-0004-5. PMID 22238004
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Stout JR, Smith-Ryan AE, Fukuda DH, Kendall KL, Moon JR, Hoffman JR, Wilson JM, Oliver JS, Mustad VA. Effect of calcium beta-hydroxy-beta-methylbutyrate (CaHMB) with and without resistance training in men and women 65+yrs: a randomized, double-blind pilot trial. Exp Gerontol. 2013 Nov;48(11):1303-10. doi: 10.1016/j.exger.2013.08.007. Epub 2013 Aug 24. PMID 23981904
- [Background] Cooper R, Hardy R, Bann D, Aihie Sayer A, Ward KA, Adams JE, Kuh D; MRC National Survey of Health and Development Scientific and Data Collection Team. Body mass index from age 15 years onwards and muscle mass, strength, and quality in early old age: findings from the MRC National Survey of Health and Development. J Gerontol A Biol Sci Med Sci. 2014 Oct;69(10):1253-9. doi: 10.1093/gerona/glu039. Epub 2014 Mar 28. PMID 24682351
- [Background] Holecek M. Beta-hydroxy-beta-methylbutyrate supplementation and skeletal muscle in healthy and muscle-wasting conditions. J Cachexia Sarcopenia Muscle. 2017 Aug;8(4):529-541. doi: 10.1002/jcsm.12208. Epub 2017 May 10. PMID 28493406
- [Background] He X, Duan Y, Yao K, Li F, Hou Y, Wu G, Yin Y. beta-Hydroxy-beta-methylbutyrate, mitochondrial biogenesis, and skeletal muscle health. Amino Acids. 2016 Mar;48(3):653-664. doi: 10.1007/s00726-015-2126-7. Epub 2015 Nov 14. PMID 26573541
- [Background] Barry BK, Carson RG. The consequences of resistance training for movement control in older adults. J Gerontol A Biol Sci Med Sci. 2004 Jul;59(7):730-54. doi: 10.1093/gerona/59.7.m730. PMID 15304540
- [Background] Liu CJ, Latham NK. Progressive resistance strength training for improving physical function in older adults. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD002759. doi: 10.1002/14651858.CD002759.pub2. PMID 19588334
- [Background] Wandrag L, Brett SJ, Frost G, Hickson M. Impact of supplementation with amino acids or their metabolites on muscle wasting in patients with critical illness or other muscle wasting illness: a systematic review. J Hum Nutr Diet. 2015 Aug;28(4):313-30. doi: 10.1111/jhn.12238. Epub 2014 May 8. PMID 24807079
- [Background] Morton RW, Murphy KT, McKellar SR, Schoenfeld BJ, Henselmans M, Helms E, Aragon AA, Devries MC, Banfield L, Krieger JW, Phillips SM. A systematic review, meta-analysis and meta-regression of the effect of protein supplementation on resistance training-induced gains in muscle mass and strength in healthy adults. Br J Sports Med. 2018 Mar;52(6):376-384. doi: 10.1136/bjsports-2017-097608. Epub 2017 Jul 11. PMID 28698222
- [Background] Bear DE, Langan A, Dimidi E, Wandrag L, Harridge SDR, Hart N, Connolly B, Whelan K. beta-Hydroxy-beta-methylbutyrate and its impact on skeletal muscle mass and physical function in clinical practice: a systematic review and meta-analysis. Am J Clin Nutr. 2019 Apr 1;109(4):1119-1132. doi: 10.1093/ajcn/nqy373. PMID 30982854
- [Background] Vukovich MD, Stubbs NB, Bohlken RM. Body composition in 70-year-old adults responds to dietary beta-hydroxy-beta-methylbutyrate similarly to that of young adults. J Nutr. 2001 Jul;131(7):2049-52. doi: 10.1093/jn/131.7.2049. PMID 11435528
- [Background] Courel-Ibanez J, Vetrovsky T, Dadova K, Pallares JG, Steffl M. Health Benefits of beta-Hydroxy-beta-Methylbutyrate (HMB) Supplementation in Addition to Physical Exercise in Older Adults: A Systematic Review with Meta-Analysis. Nutrients. 2019 Sep 3;11(9):2082. doi: 10.3390/nu11092082. PMID 31484462
- [Background] Rangel Peniche DB, Raya Giorguli G, Aleman-Mateo H. Accuracy of a predictive bioelectrical impedance analysis equation for estimating appendicular skeletal muscle mass in a non-Caucasian sample of older people. Arch Gerontol Geriatr. 2015 Jul-Aug;61(1):39-43. doi: 10.1016/j.archger.2015.03.007. Epub 2015 Apr 1. PMID 25857600
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Sanchez-Arenas R, Vargas-Alarcon G, Sanchez-Garcia S, Garcia-Pena C, Gutierrez-Gutierrez L, Grijalva I, Garcia-Dominguez A, Juarez-Cedillo T. Value of EQ-5D in Mexican city older population with and without dementia (SADEM study). Int J Geriatr Psychiatry. 2014 May;29(5):478-88. doi: 10.1002/gps.4030. Epub 2013 Oct 3. PMID 24123291
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Nissen S, Sharp RL, Panton L, Vukovich M, Trappe S, Fuller JC Jr. beta-hydroxy-beta-methylbutyrate (HMB) supplementation in humans is safe and may decrease cardiovascular risk factors. J Nutr. 2000 Aug;130(8):1937-45. doi: 10.1093/jn/130.8.1937. PMID 10917905